CLINICAL TRIAL: NCT04368325
Title: A Correlation of Low Serum Creatinine Levels and Respiratory Function in the Mechanically Ventilated Patients in the Intensive Care Unit
Brief Title: Low Creatinine Level and Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-7
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Intensive Care Unit; Respiratory Insufficiency; Muscle Weakness
Keywords: Low serume creatinine levels, respiratory insufficiency, ICU
MeSH Terms: conditions — Respiratory Insufficiency; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Total of 46 patients with low serum creatinine levels whose values were obtained from the central laboratory with inclusion criteria (< 40mmol/L)
  Interventions: Diagnostic Test: Serum creatinine levels
- Control group: A total of 61 consecutive patients were obtained who were treated in ICU CHC Osijek, according to the date of admission.
  Interventions: Diagnostic Test: Serum creatinine levels

INTERVENTIONS:
Diagnostic Test: Serum creatinine levels — Comparison of treatment length using mechanical ventilaton, length of stay in ICU, survival between two groups

SUMMARY:
Low creatinine levels may be a sign of muscle atrophy or weakness, and therefore predictive for respiratory insufficiency in the Intensive care unit (ICU) patients. The investigators compared the outcomes of participants with low creatinine levels with subsequent ICU participants admitted into ICU in the tertiary hospital.

DETAILED DESCRIPTION:
The investigators have found a total of 46 participants with low creatinine levels and compared their outcome data with a group of participants with normal or high creatinine levels (control group, N=61). Low creatinine was defined as values of ≤40 μmol/L. Demographic data, type of admission (medical vs. surgical), hemoglobin values, CRP, and ventilator days were compared. A statistical analysis was performed using chi square and T-test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for study group was value of ≤40 µmol/L serume creatinine level during hospitalization in ICU from July 2015 to November 2016.

Exclusion Criteria:

* Patients who were younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group was selected by measuring low serume creatinine levels (≤40 µmol/L) during the treatment in ICU. Control group was obtained by consecutive selection of patients according to the date of admission to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-05-17 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Length of mechanical ventilation treatment in group with low serume creatinine level | Through study completion, an average of 1 year
  The investigators compared length of mechanical ventilation treatment between group with low serume creatinine level and control group

SECONDARY OUTCOMES:
Length of stay in ICU in group with low serume creatinine level | Through study completion, an average of 1 year
  The investigators compared length of stay in ICU between group with low serume creatinine level and control group
White blood cell values in group with low creatinine level | Through study completion, an average of 1 year
  The investigators compared white blood cell values between group with low creatinine level and control group
Hemoglobine values in group with low creatinine level | Through study completion, an average of 1 year
  The investigators compared hemoglobine values between group with low creatinine level and control group
Number of patients who started nutrition in ICU | Through study completion, an average of 1 year
  The investigators compared number of patients between group with low creatinine level and control group who started nutrition in ICU
Platelets values in group with low creatinine level | Through study completion, an average of 1 year
  The investigators compared platelet values between group with low creatinine level and control group
Number of patients who receive blood products transfusion | Through study completion, an average of 1 year
  The investigators compared number of patients who received blood products between group with low creatinine level and control group
Number of patients discharged | Through study completion, an average of 1 year
  The investigators compared number of patients who were discharged from intensive care unit to the ward between group with low creatinine level and control group

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, MD; PhD., Study Chair — Osijek University Hospital
Locations (1):
- University hospital centre Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All the data recorded will be available after the manuscript will be published, upon the request by stjepan.grga.milankovic@gmail.com
Supporting Information: Study Protocol, CSR
Time Frame: After the publication of the manuscript in the medical journal
Access Criteria: Free available to anyone

REFERENCES:
- [Background] Vo P, Kharasch VS. Respiratory failure. Pediatr Rev. 2014 Nov;35(11):476-84; quiz 485-6. doi: 10.1542/pir.35-11-476. PMID 25361907
- [Background] Briones Claudett KH. Noninvasive ventilation in the event of acute respiratory failure in patients with idiopathic pulmonary fibrosis: waiting for? J Crit Care. 2014 Dec;29(6):1128. doi: 10.1016/j.jcrc.2014.07.016. Epub 2014 Jul 22. No abstract available. PMID 25201432
- [Background] Schwabbauer N, Berg B, Blumenstock G, Haap M, Hetzel J, Riessen R. Nasal high-flow oxygen therapy in patients with hypoxic respiratory failure: effect on functional and subjective respiratory parameters compared to conventional oxygen therapy and non-invasive ventilation (NIV). BMC Anesthesiol. 2014 Aug 7;14:66. doi: 10.1186/1471-2253-14-66. eCollection 2014. PMID 25110463
- [Background] Zielinski J, MacNee W, Wedzicha J, Ambrosino N, Braghiroli A, Dolensky J, Howard P, Gorzelak K, Lahdensuo A, Strom K, Tobiasz M, Weitzenblum E. Causes of death in patients with COPD and chronic respiratory failure. Monaldi Arch Chest Dis. 1997 Feb;52(1):43-7. PMID 9151520
- [Background] Pettenuzzo T, Fan E. 2016 Year in Review: Mechanical Ventilation. Respir Care. 2017 May;62(5):629-635. doi: 10.4187/respcare.05545. PMID 28442589
- [Background] Sahetya S, Allgood S, Gay PC, Lechtzin N. Long-Term Mechanical Ventilation. Clin Chest Med. 2016 Dec;37(4):753-763. doi: 10.1016/j.ccm.2016.07.014. Epub 2016 Oct 14. PMID 27842754
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] Datta D, Foley R, Wu R, Grady J, Scalise P. Can Creatinine Height Index Predict Weaning and Survival Outcomes in Patients on Prolonged Mechanical Ventilation After Critical Illness? J Intensive Care Med. 2018 Feb;33(2):104-110. doi: 10.1177/0885066616648133. Epub 2016 May 13. PMID 27179057
- [Background] Lai YC, Ruan SY, Huang CT, Kuo PH, Yu CJ. Hemoglobin levels and weaning outcome of mechanical ventilation in difficult-to-wean patients: a retrospective cohort study. PLoS One. 2013 Aug 28;8(8):e73743. doi: 10.1371/journal.pone.0073743. eCollection 2013. PMID 24015310
- [Background] Lee JJ, Waak K, Grosse-Sundrup M, Xue F, Lee J, Chipman D, Ryan C, Bittner EA, Schmidt U, Eikermann M. Global muscle strength but not grip strength predicts mortality and length of stay in a general population in a surgical intensive care unit. Phys Ther. 2012 Dec;92(12):1546-55. doi: 10.2522/ptj.20110403. Epub 2012 Sep 13. PMID 22976446
- [Background] Ellis CS. Improving Nutrition in Mechanically Ventilated Patients. J Neurosci Nurs. 2015 Oct;47(5):263-70; quiz E1. doi: 10.1097/JNN.0000000000000161. PMID 26348431
- [Background] Coudroy R, Jamet A, Petua P, Robert R, Frat JP, Thille AW. High-flow nasal cannula oxygen therapy versus noninvasive ventilation in immunocompromised patients with acute respiratory failure: an observational cohort study. Ann Intensive Care. 2016 Dec;6(1):45. doi: 10.1186/s13613-016-0151-7. Epub 2016 May 20. PMID 27207177
- [Background] Weiler N, Waldmann J, Bartsch DK, Rolfes C, Fendrich V. Outcome in patients with long-term treatment in a surgical intensive care unit. Langenbecks Arch Surg. 2012 Aug;397(6):995-9. doi: 10.1007/s00423-012-0966-0. Epub 2012 Jun 15. PMID 22699745
- [Background] van Vught LA, Klein Klouwenberg PM, Spitoni C, Scicluna BP, Wiewel MA, Horn J, Schultz MJ, Nurnberg P, Bonten MJ, Cremer OL, van der Poll T; MARS Consortium. Incidence, Risk Factors, and Attributable Mortality of Secondary Infections in the Intensive Care Unit After Admission for Sepsis. JAMA. 2016 Apr 12;315(14):1469-79. doi: 10.1001/jama.2016.2691. PMID 26975785